CLINICAL TRIAL: NCT06828900
Title: Empowering Caregivers in ADHD Treatment Decisions: a Four-arm Randomized Controlled Trial Comparing Standard Care, a Decision Aid, Decision Coaching, and AI-driven Support
Brief Title: Empowering Caregivers in ADHD Treatment: Standard Care Vs. Decision Aid, Coaching, and AI Support
Acronym: ADHD SDM
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Ariel University (Other)
Collaborators: Tel Aviv University (Other); University of Ottawa (Other)
Responsible Party: Principal Investigator, Yulia Gendler, Principal Investigator, Head of Nursing Department, Ariel University, Israel, Ariel University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: AU-HEA-YG-20240520; RA2100000224 (Other Grant/Funding Number: Ariel University)
Record Dates: First submitted 2025-02-05; First posted 2025-02-17 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-01

CONDITIONS: ADHD; ADHD, ADD; Shared Decision Making
Keywords: ADHD; Shared decision making; Decision aids; Decision coaching; AI-driven support; ADHD medical treatment
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Decision Support Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Control (Standard Care) (Active Comparator): Participants will undergo the typical clinical consultation process for ADHD treatment decisions without additional decision support interventions. Parents will meet with a physician who will present the available treatment options, based on standard clinical guidelines. The physician will answer any questions parents may have but will not use structured decision aids, coaching, or AI-driven tools. Parents will then make a treatment decision based on this discussion. This approach reflects real-world clinical encounters where parents rely solely on physician-provided information.
  Interventions: Behavioral: Written Decision Aid; Behavioral: Decision Aid + Decision Coaching; Behavioral: AI-Driven Support
- AI-Driven Support (Active Comparator): Participants will interact with a large language model-based AI tool (Claude) to assist in their decision-making process regarding medication vs. no medication for ADHD treatment. This AI-driven intervention is designed to provide structured, personalized decision support while maintaining an unbiased, evidence-based approach.
  Participants will receive 10 structured prompts to ask the AI, covering key aspects of ADHD treatment (e.g., benefits and risks of medication, long-term outcomes, alternatives).
  Following this structured phase, participants will have 15 minutes of free interaction with the AI to explore any remaining questions or concerns.
  At the end of the session, they will receive a summary output of their AI interactions to review.
  The AI tool is designed to translate complex medical information into user-friendly language, provide comparative treatment insights, and help parents clarify their values and concerns. However, it will not offer direct medical recommendations.
  Interventions: Behavioral: Written Decision Aid; Behavioral: Decision Aid + Decision Coaching
- Decision Aid + Decision Coaching (Active Comparator): Participants will receive the written decision aid booklet, developed based on IPDAS guidelines, along with a one-on-one decision coaching session. The decision coaching will follow a structured script based on the Ottawa Personal Decision Guide (OPDG), refined through training with the principal investigator (PI). The decision coach will not give medical advice but will help parents clarify their values, address uncertainties, and weigh the benefits and risks of medication vs. no medication. Through guided value clarification exercises, parents will explore their concerns and preferences to make a well-informed decision.
  Interventions: Behavioral: Written Decision Aid; Behavioral: AI-Driven Support
- Written Decision Aid (Active Comparator): Participants will receive a structured booklet developed based on IPDAS guidelines to support informed decision-making regarding medication vs. no medication for ADHD treatment. The booklet provides a clear explanation of ADHD, the role of medication, and the option of not using medication, including the potential benefits, risks, and uncertainties of each choice. It presents evidence-based information in a balanced manner, helping parents understand possible outcomes such as symptom management, side effects, and long-term considerations. The booklet also includes value clarification exercises to help parents align their decision with personal preferences and concerns.
  Interventions: Behavioral: Decision Aid + Decision Coaching; Behavioral: AI-Driven Support

INTERVENTIONS:
Behavioral: Written Decision Aid — Participants will receive a structured booklet developed based on IPDAS guidelines to support informed decision-making regarding medication vs. no medication for ADHD treatment. The booklet provides a clear explanation of ADHD, the role of medication, and the option of not using medication, including the potential benefits, risks, and uncertainties of each choice. It presents evidence-based information in a balanced manner, helping parents understand possible outcomes such as symptom management, side effects, and long-term considerations. The booklet also includes value clarification exercises to help parents align their decision with personal preferences and concerns.
  Other Names: PtDA
  Arms: AI-Driven Support; Control (Standard Care); Decision Aid + Decision Coaching
Behavioral: Decision Aid + Decision Coaching — Participants will receive the written decision aid booklet, developed based on IPDAS guidelines, along with a one-on-one decision coaching session. The decision coaching will follow a structured script based on the Ottawa Personal Decision Guide (OPDG), refined through training with the principal investigator (PI). The decision coach will not give medical advice but will help parents clarify their values, address uncertainties, and weigh the benefits and risks of medication vs. no medication. Through guided value clarification exercises, parents will explore their concerns and preferences to make a well-informed decision.
  Arms: AI-Driven Support; Control (Standard Care); Written Decision Aid
Behavioral: AI-Driven Support — Participants will interact with a large language model-based AI tool (Claude) to assist in their decision-making process regarding medication vs. no medication for ADHD treatment. This AI-driven intervention is designed to provide structured, personalized decision support while maintaining an unbiased, evidence-based approach.
  Participants will receive 10 structured prompts to ask the AI, covering key aspects of ADHD treatment (e.g., benefits and risks of medication, long-term outcomes, alternatives).
  Following this structured phase, participants will have 15 minutes of free interaction with the AI to explore any remaining questions or concerns.
  At the end of the session, they will receive a summary output of their AI interactions to review.
  The AI tool is designed to translate complex medical information into user-friendly language, provide comparative treatment insights, and help parents clarify their values and concerns. However, it will not offer direct medical recommendations.
  Arms: Control (Standard Care); Decision Aid + Decision Coaching; Written Decision Aid

SUMMARY:
The goal of this clinical trial is to evaluate different decision-support interventions to help parents make informed treatment decisions for their children with ADHD. The study will compare four approaches to assess their impact on decision-making quality, decisional conflict, and treatment adherence among parents of children aged 6-17 years diagnosed with ADHD.

The main questions it aims to answer are:

Does providing parents with decision-support tools improve decision-making quality compared to standard care? Do decision aid, decision aid + decision coaching, and AI-driven support further enhance parental self-efficacy, knowledge, and adherence to treatment decisions?

Standard care (physician consultation only) A written decision aid (structured booklet) Decision aid + decision coaching (booklet + one-on-one coaching session) AI-driven support (interaction with an AI tool)

Participants will:

Complete a baseline questionnaire before the intervention Receive their assigned decision-support intervention (if applicable) Complete follow-up questionnaires at 2 weeks and 3 months after the intervention Report on treatment decisions and medication adherence over 3 months This study will determine whether structured decision aids, coaching, or AI-driven tools improve parental decision-making and treatment adherence in ADHD care.

DETAILED DESCRIPTION:
This randomized controlled trial (RCT) aims to evaluate the effectiveness of different decision-support interventions in helping parents of children with ADHD make informed treatment decisions. The study will assess the impact of structured decision aids, decision coaching, and AI-driven support on parental decision-making quality, decisional conflict, self-efficacy, knowledge, and treatment adherence. Participants will be randomly assigned to one of four study arms: standard care, a written decision aid, decision aid plus decision coaching, or AI-driven support. Outcomes will be measured at baseline, two weeks, and three months post-intervention.

Rationale

ADHD is a common neurodevelopmental disorder affecting children worldwide. Treatment options primarily include medication or no medication, each with associated risks and benefits. Shared Decision Making (SDM) is recognized as a best-practice model, ensuring treatment decisions align with parental values and preferences. However, parents often face challenges in weighing options, understanding treatment effects, and feeling confident in their decisions. This study seeks to compare decision-support interventions to determine their effectiveness in enhancing decision-making quality, reducing decisional conflict, and improving parental knowledge and treatment adherence.

Study Design

This is a four-arm, parallel-group, randomized controlled trial. Participants will be randomly assigned in a 1:1:1:1 ratio to one of four arms:

Standard Care (Control Group): Parents receive a routine consultation with their physician, discussing ADHD treatment options without additional structured decision-support tools.

Written Decision Aid (DA): Parents receive a structured booklet, developed using IPDAS guidelines, detailing medication vs. no medication options, including their risks and benefits, to facilitate informed decision-making.

Decision Aid + Decision Coaching (DA+DC): Parents receive the written decision aid along with a one-on-one decision coaching session, where a trained facilitator helps them clarify values, address concerns, and enhance decision confidence.

AI-Driven Support: Parents interact with an AI-based decision support tool (Claude), initially responding to 10 structured prompts, followed by 15 minutes of free interaction, and then receiving an AI-generated summary of their decision-relevant queries.

Participant Recruitment and Enrollment

Participants will be recruited through an open call from the research lab. Interested individuals will contact the research assistant, who will screen for eligibility and obtain informed consent before randomization. Upon enrollment, participants will complete a baseline questionnaire assessing their initial decision-making state, knowledge, and values. Those assigned to one of the intervention arms will receive their respective decision-support intervention immediately after completing the baseline assessment.

Interventions

Standard Care: Participants will discuss ADHD treatment options with their physician without structured decision support.

Written Decision Aid: A booklet designed based on IPDAS criteria, containing balanced, evidence-based content about medication vs. no medication, value clarification exercises, and FAQs to enhance comprehension.

Decision Coaching: A trained facilitator will conduct a structured decision coaching session, using a script developed based on the Ottawa Personal Decision Guide (OPDG). The session will help parents explore treatment preferences, clarify values, and express concerns in a structured manner.

AI-Driven Support: Parents will interact with Claude, an AI-based large language model, following structured prompts and engaging in open-ended queries to explore ADHD treatment decisions. The AI-generated summary will provide key insights and reinforce understanding.

Outcome Measures

Primary Outcomes:

Decisional Conflict (DCS): Measures parental uncertainty, clarity of values, and confidence in treatment decisions. Higher scores indicate greater uncertainty, while lower scores reflect improved decision-making clarity.

Decision-Making Quality (DMQS): Evaluates how well-informed and values-aligned the parent's decision is, reflecting their engagement in a structured, evidence-based decision-making process.

Secondary Outcomes:

Parental Knowledge (CAKe): A 10-item questionnaire assessing understanding of ADHD and treatment options.

Parents' Values: A 6-item scale measuring the importance parents assign to various treatment-related outcomes.

Health Literacy (REALM): A validated tool screening for the ability to comprehend medical information.

Numeracy (SNS): An 8-item scale assessing mathematical ability and preference for numerical information.

Decision Self-Efficacy: An 11-item scale measuring parents' confidence in making an informed treatment decision.

ADHD Care: Tracks treatment received and medication adherence over three months.

Preparation for Decision-Making: A validated scale assessing how well the decision aid prepared parents for shared decision-making.

Preference for SDM: A single-item question evaluating the parent's preferred level of involvement in decision-making.

Demographics: Age, gender, education level, nationality, religion, religiosity, marital status, and number of children.

Data Collection and Follow-Up

Baseline Assessment: Participants complete questionnaires before the intervention.

Post-Intervention Assessment: Follow-up assessments at two weeks and three months after intervention.

ADHD Care Tracking: Parents report treatment choices and adherence over the three-month period.

Sample Size and Randomization

A power analysis determined that 144 participants (36 per arm) are needed to detect a meaningful difference in decisional conflict with 80% power and a 5% significance level, accounting for a 10% dropout rate. Randomization will be conducted using computer-generated block randomization to ensure balanced distribution across arms.

Statistical Analysis Plan

Data will be analyzed using SPSS version 29 and R. Statistical methods include:

Descriptive statistics: Means, standard deviations, frequencies, and percentages for baseline characteristics.

Comparative analyses:

Paired t-tests or Wilcoxon signed-rank tests for pre-post changes.

One-way ANOVA or Kruskal-Wallis tests for subgroup comparisons.

Regression models:

Linear regression for relationships between SDM measures and continuous outcomes.

Logistic regression for categorical outcomes such as treatment adherence.

Multiple imputation methods will address missing data if the rate exceeds 5%.

Sensitivity analyses will validate the robustness of findings.

Ethical Considerations

This study has been approved by the Ariel University IRB (AU-HEA-YG-20240520). All participants will provide written informed consent before participation. Data confidentiality will be maintained through de-identified coding and secure storage.

Expected Impact

This study will provide valuable insights into the effectiveness of decision-support interventions in ADHD treatment. Findings may inform best practices for integrating decision aids, coaching, and AI-driven tools into clinical workflows, enhancing shared decision-making and improving parental confidence, treatment adherence, and child health outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Parents or legal guardians of children aged 6-17 diagnosed with ADHD.
* Able to provide informed consent.
* Willing to participate in all study activities, including follow-up assessments.

Exclusion Criteria:

* Non-Hebrew-speaking parents (due to the language-based intervention materials).
* Parents who have previously participated in ADHD decision aid trials.
* Parent of children with severe comorbid psychiatric conditions requiring urgent psychiatric care

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-11-19 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Decisional conflict | Before the intervention, 2 weeks after and 3 months after
  Decisional conflict refers to the uncertainty parents experience when making treatment decisions for their child, particularly when weighing the benefits and risks of medication versus no medication for ADHD. It reflects how informed they feel about their options, how clear they are about their values, and how supported they feel in the decision-making process. Higher decisional conflict scores indicate greater uncertainty, confusion, or lack of confidence, suggesting that parents may feel uninformed, pressured, or unsure about which option aligns best with their values and preferences. A reduction in decisional conflict over time suggests that parents have gained clarity, confidence, and a better understanding of their options, leading to a more informed and satisfactory decision. This change is a key indicator of the effectiveness of decision-support interventions in helping parents navigate ADHD treatment choices.
Decision-Making Quality | 2 weeks and 3 months after the intervention
  he Decision-Making Quality Scale (DMQS) assesses the extent to which a parent's decision is informed, aligned with their values, and consistent with SDM principles. The DMQS evaluates how thoroughly an individual considers alternatives, gathers and integrates relevant information, and deliberates before making a final choice . Higher scores on the DMQS indicate a higher-quality decision-making process, characterized by greater knowledge about the decision at hand, a more deliberate weighing of risks and benefits, and stronger alignment between the chosen option and the individual's values. Conversely, lower scores suggest a decision that is less informed, potentially rushed, or influenced by external pressures rather than a systematic evaluation of options
  . This measure is crucial in ADHD treatment decision-making, as it captures the degree to which parents engage in a thoughtful and well-supported choice regarding their child's care.

SECONDARY OUTCOMES:
Knowledge | Before the intervention, 2 weeks after and 3 months after
  Knowledge questionnaire consists of ten structured questions, each designed to assess a specific aspect of ADHD knowledge, including its symptoms, causes, treatment mechanisms, and long-term management strategies. Participants will respond using a three-option format: 'true', 'false', or 'don't know'. Higher scores indicate a greater understanding of ADHD and its treatments, while lower scores may reflect misconceptions or a lack of essential knowledge that could impact decision-making quality. Knowledge scores will be analyzed both as a continuous variable and categorized into low, moderate, and high knowledge levels to assess how well each intervention supports parental learning.
Parents' values | 2 weeks and 3 months after the intervention
  Assessed through six structured questions designed to evaluate the relative importance parents place on different aspects of their child's well-being, academic performance, and overall functioning. An example question includes: "How important is it to you that your child is able to concentrate during classes at school?" Each question is rated on a six-point Likert scale ranging from 0 ('not important') to 5 ('very important'), allowing for a nuanced understanding of how strongly parents prioritize specific treatment outcomes. Higher scores reflect stronger preferences for symptom management through medical intervention, while lower scores may indicate a greater openness to non-medication approaches or a focus on other aspects of the child's development.
Health literacy | Before the intervention
  Health literacy is a crucial factor influencing how well parents understand medical information, weigh treatment options, and engage in shared decision-making (SDM). In this study, parental health literacy will be assessed using the Rapid Estimate of Adult Literacy in Medicine (REALM) questionnaire, a validated tool designed to identify individuals with inadequate health literacy. The REALM consists of three brief, structured questions, which have been validated to screen for difficulties in reading and comprehending medical information.
Numeracy | Before the intervention
  Numeracy will be assessed using the Subjective Numeracy Scale (SNS), an 8-item self-report measure evaluating both perceived mathematical ability and preference for numerical versus prose-based information. The scale consists of two subscales: one measuring confidence in performing mathematical tasks (e.g., calculating percentages, understanding probabilities) and the other assessing preference for receiving information in numerical versus verbal formats. Each item is rated on a Likert scale, with higher scores indicating greater numeracy skills and a stronger preference for numerical data. Lower scores suggest a need for simplified, prose-based explanations, which may influence how parents process ADHD treatment information.
Decision self efficacy | Before the intervention, 2 weeks and 3 months after
  Decision self-efficacy will be assessed using an 11-item questionnaire designed to measure a parent's confidence in their ability to make an informed treatment decision for their child. The scale evaluates key aspects of decision-making, including gathering necessary information, asking relevant questions, expressing opinions, and considering available options. Each item is rated on a 5-point Likert scale ranging from 0 ("not at all confident") to 4 ("extremely confident"), with higher scores indicating greater self-efficacy in navigating the decision-making process.
  This measure captures how well parents feel equipped to engage in shared decision-making (SDM), advocate for their child's needs, and communicate effectively with healthcare providers. Higher scores suggest greater confidence in actively participating in treatment decisions, while lower scores may indicate uncertainty or hesitation in the decision-making process.
ADHD care | 3 months after the intervention
  ADHD care will be assessed by tracking the type of treatment received and medication adherence over the three months following the intervention. Parents will report whether their child started, continued, or discontinued medication, as well as any changes in treatment plans, including switching medications or adjusting dosages. Additionally, adherence to pharmacological treatment will be measured by recording the number of days the child took the prescribed medication within the follow-up period.
Preparation for decision-making | Before the intervention, 2 weeks after the intervention
  reparation for decision-making will be assessed using a validated scale designed to measure how well participants perceive the decision aid's usefulness in helping them prepare for discussions with clinicians and engage in Shared Decision Making (SDM). This scale evaluates key aspects such as whether the decision aid helped clarify treatment options, increased confidence in discussing concerns, and facilitated communication with healthcare providers.
  Participants will respond using a 5-point Likert scale ranging from 1 ("not at all") to 5 ("a great deal"), with higher scores indicating a stronger belief that the decision aid was effective in preparing them for informed discussions and active participation in SDM.
Preference for SDM | 2 weeksf after the intervention
  Preference for Shared Decision-Making (SDM) will be assessed using a single-item question that captures how participants prefer to engage in the ADHD treatment decision-making process. This question evaluates the extent to which parents want to collaborate with their child's physician in making the final treatment choice.
  Participants will select one of five response options, ranging from a fully physician-led decision to a fully patient-led decision:
  My doctor will make the decision with little input from me. My doctor will make the decision but will seriously consider my opinion. My doctor and I will make the decision together. I will make the decision after seriously considering my doctor's opinion. I will make the decision with little input from my doctor. This measure provides insight into how much control parents wish to have in the decision-making process and whether this preference shifts after exposure to decision-support interventions.
Demographics | Before the intervention
  Demographic data will be collected to characterize the study population and explore potential influences on ADHD treatment decision-making. Participants will self-report their:
  Age (in years) Gender (male, female, non-binary/prefer not to say) Education level (primary, secondary, diploma, academic degree) Nationality Religion (Jewish, Muslim, Christian, Druze, other) Religiosity (secular, traditional, religious, ultra-Orthodox) Marital status (single, married, divorced, widowed) Number of children

CONTACTS AND LOCATIONS:
Overall Officials: Yulia Gendler, PhD, Principal Investigator — 'MyHealthAid' research lab - Ariel University
Locations (1):
- Ariel University, Ariel, Israel, Israel

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) supporting the findings of this study will be made available upon reasonable request. Data will be accessible to qualified researchers affiliated with academic or non-profit institutions, subject to approval. Requests should be submitted to yuliage@ariel.ac.il. Data will be stored in Open Science Framework (OSF) to ensure secure and long-term access. The dataset will be available for 5 years post-publication. Researchers must agree to a data use agreement (DUA) specifying ethical usage, proper citation, and compliance with institutional review board (IRB) requirements for secondary use.